CLINICAL TRIAL: NCT06809088
Title: Comparison of Safety and Efficacy of Tailored Versus Fixed Dose Albumin for the Management of Patients With Cirrhosis and Sepsis Associated Acute Kidney Injury - A Randomised Control Trial
Brief Title: Comparison of Safety and Efficacy of Tailored Versus Fixed Dose Albumin for the Management of Patients With Cirrhosis and Sepsis Associated Acute Kidney Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-AKI-04
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Liver Cirrhosis; Acute Kidney Injury
MeSH Terms: conditions — Liver Cirrhosis; Acute Kidney Injury | interventions — Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Regimen (Experimental): * 25% albumin infusion with monitoring of
  * Hrly - MAP, HR, Urine output, Respiratory rate,SpO2 ,Temperature
  * 3Hrly - POCUS, IVC Target <20 with respiratory phase variability, Lung USG with absence of B lines ,
  * Daily - S.Cr, eGFR, Chest Xray, 2D Echo,Renal Resistive Index
  Interventions: Biological: Albumin
- Standard medical therapy (Active Comparator): As defined in Revised consensus of International Club of Ascites and ADQI for AKI resolution Dosing of Albumin to be kept at 1gm/KG body weight daily
  * Hrly - MAP, HR, Urine output, Respiratory rate,SpO2 ,Temperature
  * 3Hrly - POCUS, IVC Target <20 with respiratory phase variability, Lung USG with absence of B lines ,
  * Daily - S.Cr, eGFR, Chest Xray, 2D Echo,Renal Resistive Index, SOFA scoring
  Interventions: Other: Standard Medical Treatment

INTERVENTIONS:
Biological: Albumin — Albumin
  Arms: Personalized Regimen
Other: Standard Medical Treatment — Standard Medical Treatment
  Arms: Standard medical therapy

SUMMARY:
Acute kidney injury accompanies about 20% of hospitalized patients with cirrhosis and in about 40% of those admitted to ICU.A critically ill patient with cirrhosis refers to an individual who has advanced liver disease (cirrhosis) and is experiencing severe and potentially life-threatening complications that require intensive medical care and monitoring. These complications might include hepatic encephalopathy, acute liver failure, severe bleeding due to portal hypertension, or other organ failures. Such patients often require specialized medical attention and interventions to stabilize their condition. The short-term prognosis of cirrhotic patients with acute kidney injury is poor, with a mortality rate higher than 65% in patients with RRT requirement. Patients with cirrhosis are prone to develop AKI . HRS comprises specific form of AKI[HRS-AKI] in patients with advanced cirrhosis and ascites, carries a high mortality risk. Role of albumin as colloid serves both as volume supplement and also as additive to vasoconstrictors. Ascites, elevated bilirubin, spontaneous bacterial peritonitis [SBP] and use of amino glycosides antibiotics had previously been identified as significant risk factors for renal failure in cirrhotic patients. The causes of AKI in cirrhotic patients include HRS [most common], others include ATN [associated mostly with sepsis]and hypovolemic shock. Three month survival ranged from 73% in patients with parenchymatous AKI to 15% for HRS. As per 2023 joint meeting of ICA and ADQI ,based on baseline serum creatinine[sCr](a lowest value obtained within the previous 3 months),AKI is defined by an absolute increases of sCr>=0.3mg/dl within 48hr or a percentage increase of sCr>=50% from baseline within 7 days and urine output <= 0.5ml/kg for >=6hrs.As per KDIGO ,three stages of AKI are defined :Stage 1]when the previous criteria are met [a relative increase of sCr 1.5-2.0from baseline, stage 2]when increase in sCr is >2folds to 3 folds from baseline and Stage 3]when there is an increase of sCr>3 folds from baseline or sCr is >4.0mg/dl with an acute increase of >0.3mg/dl or initiation of RRT. So, the study aims to analyze the role of albumin as a volume supplement and as a vasoconstrictor as well as its immunomodulatory effect in sepsis to help in resolution of AKI.Here we compare the effectiveness of personalized-dose albumin administration with fixed-dose albumin for treating acute kidney injury in patients with cirrhosis and sepsis associated AKI.

DETAILED DESCRIPTION:
Study population:

• Age - 18-70 years

Study design: Monocentric open label randomised controlled study. The study will be conducted in Department of Hepatology ILBS.

Primary Objective : Effect of personalized dose of albumin compared to fixed dose protocol in improving AKI resolution at 48 hrs.

Secondary objectives:

* To study the cumulative dose of albumin in both groups.
* Time to AKI resolution and initiation of vasoconstrictors in both the groups
* Incidence of cardiopulmonary complications in both groups
* Impact of dose of albumin on cardiac function [including CVP and IVC], intraabdominal pressure and renal perfusion [assessed by renal artery resistive index] in both groups at 24 hr and 48 hrs.
* To study the role of intraabdominal pressure, Lung USG , biomarkers of cardiac dysfunction [NT Pro BNP, Troponin T] in predicting the development of cardiopulmonary complications and AKI outcomes.
* To study the duration of AKI and need of dialysis in both groups.
* 28-day mortality in both groups

Stopping Rule:

1. With the development of cardiorespiratory adverse effects

   1. Increase in Heart rate > 10 from basal value
   2. Increase in RR > 20/min
   3. Temp > 1000 F
   4. SpO2 < 96%
   5. B lines in Lung USG
   6. IVC >= 20 with collapsibility <50% or distensibilty <18%
2. Development of allergy
3. On worsening shock ,if Noradrenaline requirement increases >0.1mcg/kg bw/min
4. worsening AKI with a]decrease in urine output b]Need of Terlipressin c]Start of RRT
5. If Downstaging of AKI does not occur on 48hr of Albumin infusion then based on GFR and urine output decision to add vasoconstrictor to be taken

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 and <70
2. patients with cirrhosis and AKI with sepsis.

Exclusion Criteria:

1. AKI- secondary to post renal causes such as nephrolithiasis
2. Patient already on maintenance hemodialysis/RRT
3. Patients with shock requiring vasopressors
4. Patient with history of structural heart disease and LVEF < 50%
5. Patient with known COPD
6. Patient on Mechanical ventilation with P/F ratio <200
7. Patient with POCUS based features of volume overload[Presence of B lines ]
8. HCC - Beyond MILAN criteria
9. Patient in need of surgical intervention
10. Patient with history of adverse reaction to Albumin infusion
11. Pregnant or Lactating Women
12. Portal or hepatic vein thrombosis
13. Volume Overload with baseline IVC >20
14. Failure to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients having resolution of AKI at 48hrs or 7days without the development of adverse events | 48hrs/7days

SECONDARY OUTCOMES:
Cumulative dose of albumin (in g/day) used in both arms at 48 hours and day 7 | 48 hours and day 7
Time to initiation of vasoconstrictors and resolution of AKI | 7 days
Proportion of patients requiring invasive or non-invasive mechanical ventilation at 48 hours and at day7 | 48 hours and day 7
Proportion of patients developing cardiopulmonary complications in both groups | 7 days
28-day mortality of hospitalized patients with AKI in Cirrhosis | 28 days
Proportion of patients with AKI progression or requiring dialysis at 48 hours and day 7 | 48 hours and day 7
SOFA score changes at 48 hrs and 7 days | 48 hours and day 7
SIRS score changes at 48 hrs and 7 days | 48 hours and day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided